CLINICAL TRIAL: NCT02111616
Title: Improving Survivorship Care Through Enhanced Communication and Coordination: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UNC HENC LCCC 1325
Record Dates: First submitted 2014-01-10; First posted 2014-04-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: cancer survivorship care; provider communication; provider care coordination
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SCP) (Active Comparator): Patient will attend a transition visit at the conclusion of cancer treatment. Patient will receive an individualized cancer survivorship care plan based on their cancer type and treatment.
  Interventions: Behavioral: Survivorship Care Plan (SCP)
- Intervention Arm (SCP + PCP visit) (Experimental): Patient will attend a transition visit at the conclusion of cancer treatment. Patient will receive an individualized cancer survivorship care plan based on their cancer type and treatment.
  SCP plus Coordinated PCP Visit: Care coordinators will schedule patient appointment with PCP within 4 weeks of treatment.
  Interventions: Behavioral: Survivorship Care Plan (SCP); Behavioral: Coordinated PCP visit

INTERVENTIONS:
Behavioral: Survivorship Care Plan (SCP) — Cancer Survivorship Care Plan (SCP) adapted from JourneyForward template. Each SCP is individualized to patient's care regimen. SCP is delivered at the conclusion of cancer treatment and during the patient's transition visit with nurse practitioner or physician assistant.
Behavioral: Coordinated PCP visit — Visit with PCP scheduled on behalf of patient at the conclusion of cancer treatment and patient's transition visit.
  Arms: Intervention Arm (SCP + PCP visit)

SUMMARY:
Purpose: Cancer survivorship is a high clinical and research priority both nationally and at the University of North Carolina. The investigators propose a randomized pilot study testing the development, implementation and evaluation of a parallel patient and streamlined provider version of a personalized Survivorship Care Plan (SCP) with lung cancer patients.

Participants: 60 lung cancer patients at Rex Cancer Center.

Procedures (methods): Participants will be recruited and randomized to the standard of care (30 patients) or intervention (30 patients) arm. Patients randomized to standard of care will receive a tailored survivorship care plan at the end of cancer treatment. Patients randomized to the intervention will receive a care plan and coordinating visit with their primary care provider. Patients will be invited to complete baseline and follow-up assessments regarding care needs and confidence in post cancer care.

All patient primary care providers will receive condensed provider versions of the care plan. Providers will be asked to evaluate how the SCP and coordinated care visit (intervention only) facilitated communication and coordination of care.

DETAILED DESCRIPTION:
Eligible participants ending or recently ending treatment will be identified weekly by the Rex Care Coordinator. The Rex Care Coordinator will contact eligible patients before cancer treatment ends to schedule an exit interview and to describe the study, get permission to share contact information with the program manager (PM), and provide the written consent form to the patient.

Two weeks prior to the scheduled exit interview, the PM will contact the patient to provide additional details about the study and obtain consent from the patient. The PM will mail baseline data collection measures to the patient to complete and bring to exit interview visit.

The PM will contact the PCP of consented patients via email or letter informing them of their patient's participation in the study and inviting them to participate as well. Providers will receive a fact sheet about the study and a confidential email link to Qualtrics to complete surveys regarding patient survivorship care. Their participation in the survey will convey consent. The link will confirm provider name and that patient is seen by the provider. A separate link will allow the provider to enter responses and maintain separation of patient identifiers and responses.

It is possible that PCPs may see multiple patients in our study, but this will not be the majority of PCPs. Providers will be asked to complete a survey for each patient. It is also possible providers may treat patients who are randomized to both arms. Because of the small sample size and the focus on feasibility, we will not limit PCPs to only see survivors in one group. The rate of this occurrence and preliminary data obtained from this pilot study will inform design/sample size calculations for the Phase III trial.

At least one week prior to the scheduled exit interview, the Rex Research Nurse will be informed by the PM to develop the SCP using the JourneyForward™ template. The Rex Research Nurse will keep a log of how long it takes to complete the SCP and any issues that arise preparing them. Tailored SCPs will be developed for each eligible patient using the template based on information on the patient's medical and cancer records.

When the patient comes to their post-treatment exit interview, their baseline surveys will be collected. Patients will receive a printed copy of their SCP during the post-treatment exit interview with the oncology nurse navigator, nurse practitioner or physician assistant. This visit will include a review of the SCP and any questions or concerns the patient may have. The PM will then randomize the patient, stratified by tumor type, to the standard of care arm (SCP alone) or the coordinated care visit arm (SCP + PCP visit).

Standard of Care Arm:

The patient's PCP will receive an abbreviated copy of the tailored SCP electronically (if accessible within the Electronic Medical Record (EMR)) or by mail. This abbreviated version contains the same treatment summary but a more concise care plan. No attempt to influence regularly scheduled appointments will be made but we will document if a visit does occur within the study window and the reason for it from patient's self-report.

Intervention Arm:

Patients randomized to the coordinated care visit arm will also have an appointment scheduled with their PCP by the research nurse within 4 weeks of the exit interview to review and discuss survivorship care. The patient's PCP will receive a copy of the abbreviated SCP electronically (if accessible within the EMR) or by mail along with suggested talking points about role clarity about what type of care the PCP will provide and when the patient should contact the PCP or their oncologist.

At six weeks following the exit interview (two weeks after the visit to the PCP for the intervention group), the PM will contact all patients to complete the follow-up measures by mail or by phone. Six weeks following the exit interview, all patients' PCPs will be contacted via phone to complete the provider measures.

ELIGIBILITY:
Inclusion Criteria:

* >21 years
* Able to read and speak English will be eligible to participate
* Diagnosed with a smoking-related cancer (initial accrual priority is lung cancer, followed by head and neck, esophageal and cervical cancer)
* Treated at Rex Cancer Center for cancer
* Completed treatment within the past three months-
* Have a designated primary care provider (PCP)

Exclusion Criteria:

* patient does not meet inclusion criteria
* patient diagnosed with metastatic cancer

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with increased patient confidence about Survivorship Care | Up to six weeks
  To compare the change in confidence about survivorship care between patients who receive a coordinated care visit with their PCP (intervention group) compared to those who do not have this visit (control group). The project will use 8 questionnaires to assess changes in patient and provider confidence and patient concerns over the course of the study. The primary objective in this one year study is to compare changes in Confidence in Survivorship Information Questionnaire (CSI) scores among patients receiving the proposed standard of care survivorship care plan (30 patients) to patients receiving care plans and a coordinated PCP visit (30 patients) to determine whether the delivery of tailored SCPs increases the confidence of survivors in receiving post treatment cancer care.

SECONDARY OUTCOMES:
Patient Activation Score | Up to 6 weeks
  To compare changes in survivor concerns, activation, perspective on care coordination, expectations and satisfaction between intervention and control group as measured by Patient Activation Measure (PAM).
Number of providers with increased confidence about survivorship | Up to 6 weeks
  To compare the change in confidence about survivorship care between PCPs who were 1) only assigned survivors in the control group, 2) only assigned survivor in the coordinated care visit and 3) who were assigned both types of survivors. This information will be captured via questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah K. Mayer, PhD, RN, Principal Investigator — University of North Carolina, Chapel Hill; Donald L Rosenstein, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Rex Cancer Center, Raleigh, North Carolina, United States

REFERENCES:
- See also: Journey Forward is a program for healthcare providers and patients who have recently completed active treatment for cancer. — http://www.journeyforward.org